CLINICAL TRIAL: NCT04522427
Title: Study of Presbyopia-correcting Intraocular Lenses in Eyes With Previous Corneal Laser Refractive Surgery
Brief Title: Study of Presbyopia-correcting Intraocular Lenses in Eyes With Previous Corneal Refractive Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Yinghong Ji
Record Dates: First submitted 2020-08-16; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Cataract; Presbyopia
Keywords: Post-corneal Refractive Surgery; Presbyopia-correcting IOL; Cataract; Efficiency; Safety
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multifocal and Extended Depth-of-Focus intraocular lenses (Experimental): Patients suffering from cataract getting phacoemulsification and Intraocular lenses(IOLs) implantation
  Interventions: Device: Use Multifocal and Extended Depth-of-Focus Intraocular Lenses(IOLs)
- Monofocal intraocular Lenses (Active Comparator): Patients suffering from cataract getting phacoemulsification and Intraocular lenses(IOLs) implantation
  Interventions: Device: Use Monofocal intraocular lenses(IOLs)

INTERVENTIONS:
Device: Use Multifocal and Extended Depth-of-Focus Intraocular Lenses(IOLs) — IOLs include AT LISA tri 839MP, AcrySof IQ PanOptix IOL, TECNIS Symfony EDOF
  Arms: Multifocal and Extended Depth-of-Focus intraocular lenses
Device: Use Monofocal intraocular lenses(IOLs) — Monofocal IOLs include 409(Zeiss), AcrySof, TECNIS IOLS
  Arms: Monofocal intraocular Lenses

SUMMARY:
This is a single-center, randomized, open, positive product, parallel controlled trial to evaluate the clinical outcomes of presbyopia-correcting intraocular lenses(IOLs) in eyes with previous corneal refractive surgery.

Specific Aim 1 (Primary): To compare the surgical successful rate of Multifocal and Extended Depth-of-Focus IOLs with Monofocal IOLs for the treatment in eyes with previous corneal refractive surgery.

Specific Aim 2 (Secondary): To study the suboptimal surgical outcomes between Multifocal and Extended Depth-of-Focus IOLs with Monofocal IOLs for the treatment in eyes with previous corneal refractive surgery.

DETAILED DESCRIPTION:
Recently, the demands for myopia correction and corneal refractive laser surgery are rising with the increased prevalence of myopia. Corneal laser refractive surgery includes photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), laser-assisted subepithelial keratomileusis ( LASEK), femtosecond assisted laser in situ keratomileusis (FS-LASIK), and small incision lenticule extraction(SMILE). At present, FS-LASIK and SMILE are the mainstream methods for correcting myopia refractive surgery with advantages of safety, reliability, predictability and stability compared with other types of refractive surgery. Cataract is the most important cause of blindness in my country and even in the world. More than 50% of blind people are caused by cataract. Many patients who have undergone corneal laser refractive surgery may develop presbyopia or cataracts with age. Phacoemulsification and intraocular lens(IOLs) implantation are the main methods for cataract due to lacking effective pharmaceutical treatments. In addition, the patients who use traditional monofocal IOLs without the ability of accommodation may fail to get rid of glasses. Therefore, a solution that can provide both distance vision and near vision is needed to the presbyopia or cataracts patients with previous corneal refractive surgery and accustomed to taking glasses off.The application of presbyopic IOL in cataract after corneal refractive surgery become extensive with the IOL technology continuously advancing, including Extended Depth-of-Focus(EDOF) IOL, multifocal IOL(especially trifocal IOL) and so on, which can improve the distance, middle, and near visual acuity conducing to reduce the rate of wearing glasses after cataract surgery.

This project is a single-center, randomized, open, positive product, parallel controlled trial to study the clinical outcomes and applied value of presbyopic IOLs, including EDOF and trifocal IOLs after corneal laser refractive surgery complicated with cataracts, and seek better solutions to enable patients to achieve satisfactory visual quality and refractive results after surgery, culminating in completing patients' demand of taking glasses off.

ELIGIBILITY:
Inclusion Criteria:

* The operated eye has ever undergone corneal refractive surgery, including PRK, LASIK, LASEK, FS-LASIK, SMILE and excluding RK
* At least one eye suffering from cataract and expected to undergo phacoemulsification and IOL implantation and cataract nuclei rigidity in the operated eye from 1 to 3 degree
* Expected to use intraocular lens power in -10.0D~+30.0D
* Willing and able to comply with scheduled visits and other study procedures.
* The need to decrease the dependence of glasses
* Signing an informed consent form

Exclusion Criteria:

* Any vision-limiting problems (e.g., corneal, retinal, infection) which could potentially limit their post-operative visual potential
* Any newly acquired ocular condition or pathology (e.g., ARMD, epiretinal membrane, chronic dry eye, irregular astigmatism, diabetic retinopathy)
* The density of corneal endothelial cells is lower than 2000/mm2
* The natural diameter of the pupil under the darkroom is less than 3mm or greater than 5.5mm
* The Kappa or Alpha angle of the operated eye is greater than 0.5mm, or the Kappa angle is greater than half of the diameter of the central refractive optical zone in the multifocal intraocular lens
* Patients with expected best corrected distance visual acuity(BCDVA) less than 0.5 (decimal vision)
* Occurrence of irregular corneal astigmatism that affects postoperative vision
* Intraocular conventional surgery within the past three months or intraocular laser surgery within one month in the operated eye
* Pregnant, lactation or planning to become pregnant in the near future
* Any surgical contraindications
* Uncontrolled systemic or ocular disease
* Use of any systemic or topical drug known to interfere with visual performance
* Other ocular surgery at the time of the cataract extraction
* Traumatic cataract or congenital bilateral cataract in the operated eye
* Getting used to reading with glasses
* High requirements for visual functions in patients' career or daily life
* Professional drivers or frequent outdoor workers at night
* A medical history of photophobia
* Amblyopia
* Excessive vision expectations after surgery or too sensitive, nervous, depressed or picky
* Unsupervised or unable to comply with scheduled visits
* The contralateral eye was judged to lose visual function
* Other situations where the researcher judges that the patient is not suitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative UDVA measured with standard visual acuity charts | Measured 3 months after cataract surgery
  postoperative uncorrected distance visual acuity(UDVA)
Postoperative UIVA measured with standard visual acuity charts | Measured 3 months after cataract surgery
  Postoperative uncorrected intermediate visual acuity(UIVA)
Postoperative UNVA measured with standard visual acuity charts | Measured 3 months after cataract surgery
  Postoperative uncorrected near visual acuity(UNVA)

SECONDARY OUTCOMES:
monocular vision measured with standard visual acuity charts | Measured first day, first week, first month, 3 months, and 6 months after cataract surgery
  Uncorrected distance visual acuity and best corrected distance visual acuity
monocular vision measured with standard visual acuity charts | Measured 1 month, 3 months, and 6 months after cataract surgery
  Uncorrected intermediate visual acuity, best corrected intermediate visual acuity, distance-corrected intermediate visual acuity, uncorrected near visual acuity, best corrected near visual acuity, and distance-corrected near visual acuity
Diopter measured by Phorometer | Measured 1 month, 3 months, and 6 months after cataract surgery
  Important factor affecting the improvement of postoperative visual function
IOL rotation stability | Measured first day, first week, first month, 3 months, and 6 months after cataract surgery
  The change in axis position will be evaluated with respect to the baseline measurement at the end of surgery. Differences in axis position will be described as rotation in degrees (0 to 360°)
Wavefront aberration measured with the iTrace (Tracey Technologies, Houston, TX) | Measured 1 month, 3 months, and 6 months after cataract surgery
  total aberration, total low-order aberration, and total high-order aberration
Contrast sensitivity measured by FACT chart | Measured 6 months after cataract surgery
  Provide accurate and comprehensive objective basis for the evaluation of visual function of cataract patients
Binocular vision measured with standard visual acuity charts | Measured 6 months after cataract surgery
  Uncorrected distance visual acuity, best corrected distance visual acuity, uncorrected intermediate visual acuity, best corrected intermediate visual acuity, distance-corrected intermediate visual acuity, uncorrected near visual acuity, best corrected near visual acuity, and distance-corrected near visual acuity.
The rate of IOL dislocation | Measured 6 months after cataract surgery
  Effectiveness evaluation index
Defocus Curve | Measured 6 months after cataract surgery
  Drawing Defocus Curve after taking the average of the data collected in each group of patients
Postoperative satisfaction：Chinese version visual function index-12(VF-12-CN) | Measured 6 months after cataract surgery
  Questionnaire survey on patients' quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Yinghong Ji, phD, Principal Investigator — Eye Institute, Eye & ENT Hospital of Fudan University
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wen D, McAlinden C, Flitcroft I, Tu R, Wang Q, Alio J, Marshall J, Huang Y, Song B, Hu L, Zhao Y, Zhu S, Gao R, Bao F, Yu A, Yu Y, Lian H, Huang J. Postoperative Efficacy, Predictability, Safety, and Visual Quality of Laser Corneal Refractive Surgery: A Network Meta-analysis. Am J Ophthalmol. 2017 Jun;178:65-78. doi: 10.1016/j.ajo.2017.03.013. Epub 2017 Mar 20. PMID 28336402
- [Background] Li M, Li M, Chen Y, Miao H, Yang D, Ni K, Zhou X. Five-year results of small incision lenticule extraction (SMILE) and femtosecond laser LASIK (FS-LASIK) for myopia. Acta Ophthalmol. 2019 May;97(3):e373-e380. doi: 10.1111/aos.14017. Epub 2019 Jan 11. PMID 30632671
- [Background] Bourne RR, Stevens GA, White RA, Smith JL, Flaxman SR, Price H, Jonas JB, Keeffe J, Leasher J, Naidoo K, Pesudovs K, Resnikoff S, Taylor HR; Vision Loss Expert Group. Causes of vision loss worldwide, 1990-2010: a systematic analysis. Lancet Glob Health. 2013 Dec;1(6):e339-49. doi: 10.1016/S2214-109X(13)70113-X. Epub 2013 Nov 11. PMID 25104599
- [Background] Tang Y, Wang X, Wang J, Huang W, Gao Y, Luo Y, Lu Y. Prevalence and Causes of Visual Impairment in a Chinese Adult Population: The Taizhou Eye Study. Ophthalmology. 2015 Jul;122(7):1480-8. doi: 10.1016/j.ophtha.2015.03.022. Epub 2015 May 16. PMID 25986897
- [Background] Keates RH, Pearce JL, Schneider RT. Clinical results of the multifocal lens. J Cataract Refract Surg. 1987 Sep;13(5):557-60. doi: 10.1016/s0886-3350(87)80114-1. PMID 3312575
- [Background] Seitz B, Langenbucher A, Nguyen NX, Kus MM, Kuchle M. Underestimation of intraocular lens power for cataract surgery after myopic photorefractive keratectomy. Ophthalmology. 1999 Apr;106(4):693-702. doi: 10.1016/S0161-6420(99)90153-7. PMID 10201589
- [Background] Chan TC, Liu D, Yu M, Jhanji V. Longitudinal evaluation of posterior corneal elevation after laser refractive surgery using swept-source optical coherence tomography. Ophthalmology. 2015 Apr;122(4):687-92. doi: 10.1016/j.ophtha.2014.10.011. Epub 2014 Dec 6. PMID 25487425
- [Background] Wang L, Hill WE, Koch DD. Evaluation of intraocular lens power prediction methods using the American Society of Cataract and Refractive Surgeons Post-Keratorefractive Intraocular Lens Power Calculator. J Cataract Refract Surg. 2010 Sep;36(9):1466-73. doi: 10.1016/j.jcrs.2010.03.044. PMID 20692556
- [Background] Ferreira TB, Pinheiro J, Zabala L, Ribeiro FJ. Comparative analysis of clinical outcomes of a monofocal and an extended-range-of-vision intraocular lens in eyes with previous myopic laser in situ keratomileusis. J Cataract Refract Surg. 2018 Feb;44(2):149-155. doi: 10.1016/j.jcrs.2017.11.007. Epub 2018 Mar 8. PMID 29526338
- [Background] Alio JL, Abdelghany AA, Abdou AA, Maldonado MJ. Cataract surgery on the previous corneal refractive surgery patient. Surv Ophthalmol. 2016 Nov-Dec;61(6):769-777. doi: 10.1016/j.survophthal.2016.07.001. Epub 2016 Jul 15. PMID 27423631
- [Background] Naseri A, McLeod SD. Cataract surgery after refractive surgery. Curr Opin Ophthalmol. 2010 Jan;21(1):35-8. doi: 10.1097/ICU.0b013e328333e9ab. PMID 19996749
- [Background] Gimbel H, Sun R, Kaye GB. Refractive error in cataract surgery after previous refractive surgery. J Cataract Refract Surg. 2000 Jan;26(1):142-4. doi: 10.1016/s0886-3350(99)00327-2. PMID 10646161
- [Background] Koch DD, Wang L. Calculating IOL power in eyes that have had refractive surgery. J Cataract Refract Surg. 2003 Nov;29(11):2039-42. doi: 10.1016/j.jcrs.2003.10.009. No abstract available. PMID 14670401
- [Background] Aramberri J. Intraocular lens power calculation after corneal refractive surgery: double-K method. J Cataract Refract Surg. 2003 Nov;29(11):2063-8. doi: 10.1016/s0886-3350(03)00957-x. PMID 14670413
- [Background] Tang M, Li Y, Huang D. An intraocular lens power calculation formula based on optical coherence tomography: a pilot study. J Refract Surg. 2010 Jun;26(6):430-7. doi: 10.3928/1081597X-20090710-02. Epub 2010 Jun 17. PMID 20677729
- [Background] Abulafia A, Hill WE, Koch DD, Wang L, Barrett GD. Accuracy of the Barrett True-K formula for intraocular lens power prediction after laser in situ keratomileusis or photorefractive keratectomy for myopia. J Cataract Refract Surg. 2016 Mar;42(3):363-9. doi: 10.1016/j.jcrs.2015.11.039. Epub 2016 Mar 19. PMID 27006324
- [Background] Wang L, Tang M, Huang D, Weikert MP, Koch DD. Comparison of Newer Intraocular Lens Power Calculation Methods for Eyes after Corneal Refractive Surgery. Ophthalmology. 2015 Dec;122(12):2443-9. doi: 10.1016/j.ophtha.2015.08.037. Epub 2015 Oct 14. PMID 26459996